CLINICAL TRIAL: NCT00124436
Title: Follow up Efficacy and Safety Study of BAL4979 in the Treatment of Chronic Hand Dermatitis Refractory to Topical Treatment
Brief Title: Follow-up Efficacy and Safety of Alitretinoin in Severe Chronic Hand Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BAP00091
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hand Dermatoses
Keywords: Patients who have been enrolled in study protocol BAP089, and whose severe chronic hand dermatitis responded with mild or moderate disease, or who relapsed
MeSH Terms: conditions — Hand Dermatoses | interventions — Alitretinoin

INTERVENTIONS:
Drug: alitretinoin

SUMMARY:
Patients who have been treated in study protocol BAP089 may have responded to treatment, and subsequently relapsed to >75% of the baseline disease severity, will be investigated for response to further treatment with alitretinoin. Also, patients who have responded with mild or moderate disease will be investigated for additional treatment effect after prolongated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in protocol BAP089
* Response of severe, treatment refractory hand dermatitis with mild or moderate, or responding patients who relapsed to 75% of baseline disease

Exclusion Criteria:

* Female patients who are pregnant or who want to become pregnant
* Female patients of child bearing potential who cannot use or who will not commit to using two effective methods of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Response of chronic hand dermatitis to study treatment as assessed by Physicians Global Assessment, at week 12 or 24

SECONDARY OUTCOMES:
Patient's global assessment
Extent of disease
Time to respond
Modified total lesion symptom score
at week 12 or 24

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruzicka, MD, Principal Investigator — University of Düsseldorf, Dermatological Hospital, Germany
Locations (1):
- Thomas Ruzicka, Düsseldorf, Germany

REFERENCES:
- [Background] Ruzicka T, Larsen FG, Galewicz D, Horvath A, Coenraads PJ, Thestrup-Pedersen K, Ortonne JP, Zouboulis CC, Harsch M, Brown TC, Zultak M. Oral alitretinoin (9-cis-retinoic acid) therapy for chronic hand dermatitis in patients refractory to standard therapy: results of a randomized, double-blind, placebo-controlled, multicenter trial. Arch Dermatol. 2004 Dec;140(12):1453-9. doi: 10.1001/archderm.140.12.1453. PMID 15611422